CLINICAL TRIAL: NCT04672070
Title: A Randomised Clinical Trial to Test the Efficacy of Selective Caries Removal (SCR) Versus Pulpotomy in Preventing Pulp Necrosis and Apical Periodontitis
Brief Title: Selective Caries Removal (SCR) Versus Pulpotomy in Preventing Pulp Necrosis and Apical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSRB 2018/01360
Record Dates: First submitted 2020-03-22; First posted 2020-12-17 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-06

CONDITIONS: Dental Caries
Keywords: vital pulp therapy; selective caries removal; pulpotomy
MeSH Terms: conditions — Dental Caries | interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Study subject (tooth) will be randomized in a 1:1 allocation ratio between the two treatment groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be done to the outcomes assessors to reduce bias during radiographic healing assessment. Participants also will not be informed of which treatment they are undergoing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective Caries Removal (Active Comparator): The patient will be treated with Selective Caries Removal (SCR)
  Interventions: Other: Selective Caries Removal
- Pulpotomy (Active Comparator): The patient will be treated with full coronal Pulpotomy.
  Interventions: Other: Pulpotomy

INTERVENTIONS:
Other: Selective Caries Removal — Selective caries are removed only for secure sealing with a direct restoration, without removing deep caries next to the pulp.
  If the pulp is exposed, pulpotomy will be performed instead and the tooth will be excluded from further analysis.
  Other Names: indirect pulp capping; partial caries removal
  Arms: Selective Caries Removal
Other: Pulpotomy — Complete caries removal and excision of the coronal pulp to the level of the root canal orifices will be performed. After haemostasis, sealing with Biodentine® and restoration.
  If the pulp is not exposed after complete caries removal, the tooth will be restored without further excavation and pulp exposure. If the pulp is assessed intra-operatively to be non-vital or not amenable to pulpotomy, root canal treatment will be performed instead. In both cases, the tooth will be excluded from further analyses.
  Other Names: full pulpotomy; coronal pulpotomy
  Arms: Pulpotomy

SUMMARY:
The study design is a randomized controlled trial and up to 120 teeth, 50 in each of the 2 groups, will be enrolled from the patients at the National University Centre for Oral Health Singapore (NUCOHS) Endodontic unit.

The primary aim of this study is to compare the efficacy of selective caries removal (SCR) and pulpotomy in preventing pulp necrosis and apical periodontitis in teeth with deep dental caries radiographically extending at least 2/3 into the width of dentine, over a review period of 6 months, 1, 3, and 5 years. The secondary aim of this study is to compare the costs (tangible i.e. restorative treatment costs, and intangible i.e. number of treatment visits and time spent at clinic to complete treatment) and tooth survival in the oral cavity, between teeth treated with SCR and pulpotomy.

DETAILED DESCRIPTION:
1. Randomisation and Blinding Teeth will be randomised to receive either SCR or Pulpotomy blindly, with 50 teeth in each group. Teeth allocated to Pulpotomy that do not subsequently have caries extending deep to reach the pulp will be excluded from the Study. Recruitment will continue until the target sample size in each group is attained , up to a maximum of 120 teeth (surplus to account for teeth that are not able to complete the allocated treatment).

   Investigators trained in SCR and Pulpotomy will perform both treatment procedures.

   For patients with multiple teeth with deep carious lesions suitable for this study, the unit of randomisation will be the individual tooth and not the patient. If it is not possible to perform treatment on all the teeth in the same visit, the operator will start on the tooth which displays the deepest lesion measured radiographically and according to clinically exigencies.

   In the event of emergency/unscheduled return visits due to pain, the patient's treatment notes will be made available to the attending dentist and emergency treatment rendered as appropriate (e.g. root canal treatment). This tooth and its relevant research data will be included as an event in the survival analysis but the tooth will be discontinued from the Trial.
2. Study Visits and Procedures Dental clinicians at National University Polyclinic (NUP) Dental Clinics and NUCOHS will follow a case selection template for patient referral. Timeframe for recruitment is up to 6months after referral to NUCOHS. The patients will be provided standard of care by their dentists according to the respective Institutional Practice, which may include Oral Health Education, Oral Health Instruction and/or scaling and polishing.

   Consent: Patients will be informed of the Study at their first visit to NUCOHS and given time to consider participation and ask questions. Written informed consent will be obtained before proceeding to Screening.

   Screening and Enrolment: Clinical and radiographic examination in line with current clinical practice to save teeth with deep caries will be conducted. When inclusion and exclusion criteria are fulfilled, the tooth will be enrolled into the study. One patient may contribute more than one tooth.

   Randomisation: This will be performed after tooth is enrolled.

   Treatment - SCR or Pulpotomy: After allocation to SCR or Pulpotomy, in both groups, interventions will be performed in a single visit under local anaesthesia and rubber dam isolation. Caries will be removed using high speed burs with water coolant starting from the periphery.

   In the SCR group, selective caries are removed only for secure sealing with a direct restoration, without removing deep caries next to the pulp.

   In the Pulpotomy group, complete caries removal and excision of the coronal pulp to the level of the root canal orifices will be performed. After haemostasis, sealing with Biodentine® and restoration.

   In either group, if the tooth is unable to complete the allocated treatment, this tooth will be excluded from the study.

   In both groups, direct restoration (e.g. composite resin or amalgam) or crowns will be provided based on remaining tooth structure, number of remaining functioning units, location of the tooth and its opposing counterpart.

   Review Appointments: Four Review visits will be conducted at the following time points:
   * 6-7 months post treatment
   * 12- 13 months post treatment
   * 36-37 months post treatment
   * 60-61 months post treatment

   Data Collection:

   Baseline data will include:
   * Relevant pain history
   * Clinical examination of the tooth, pulp and surrounding bone and mucosa
   * Routine dental radiographic examination for tooth restoration

   After treatment is completed, the following treatment data will include:
   * Time to achieve haemostasis for teeth in the pulpotomy group
   * Time taken for the procedure
   * Type of restoration placed
   * Cost of treatment
   * Cumulative time spent at the dental clinic to complete treatment

   At follow-up appointments, the review data will include:
   * Relevant pain history since the last visit
   * Clinical examination of the tooth, pulp and surrounding bone and mucosa
   * Routine dental radiographic examination to evaluate supporting bone response to the preserved pulp
   * Relevant additional procedures for teeth during review period if needed (e.g. replacement of restoration)
   * Cumulative treatment fees charged to preserve teeth (since enrolment)
   * Cumulative number of treatment visits (including any additional procedures during the review period, if any)
3. Statistical and Analytical Plans Unit of analysis is per tooth level. Descriptive analysis (mean & standard deviation and frequency and proportion, where appropriate) will be performed to summarize the baseline characteristics of recruited subjects between the two treatment groups. To study the primary objective - comparing the tooth survival without pulp pathosis between the two treatment groups at 6 months, 1 year, 3 years and 5 years, proportional z-test will be performed.

Generalized estimating equation (GEE) with binomial family distribution and log link function will be employed to study the change in tooth survival over the study follow-up period. Potential confounders and clinical predictors will be adjusted in the model.

Significance level for all statistical test is set at p-value<0.05. SPSS Statistical Package (IBM SPSS Statistics) will be used for all statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at National University Polyclinics (NUP) Dental Clinics or NUCOHS general dentistry clinics
* Aged between 21-65 years old
* Deep primary or secondary caries diagnosed on radiograph as being at least 2/3 into the thickness of dentine
* Permanent tooth with mature apices
* ASA I and II (American Society of Anesthesiologists Physical Status Classification System)
* Willing to commit to dental health education (DHE), oral hygiene instructions (OHI), restoration, and reviews of treatment completed
* Positive response to cold test with Endo-Ice® (non-lingering beyond 2 minutes) and electric pulp testing

Exclusion Criteria:

* Spontaneous and/or continuous pain associated with the carious tooth
* Pulp exposure present
* Tooth requires a post-retained core for restoration
* Tooth is required to support a fixed or removable partial denture
* Tooth with localized severe periodontitis (mobility grade ≥ 2 and/or periodontal pocket ≥ 5mm)
* Teeth with periapical lesion (defined as periapical radiolucency in connection with the apical part of the root where the width of the radiolucent lesion exceeds twice the width of the periodontal ligament space)
* Tooth needs to be extracted
* Tooth with occlusal trauma or occlusal overload (e.g. denture abutment tooth)
* Tooth is unable to complete allocated treatment
* Self-declared pregnancy
* Patient is unable to give consent (e.g. cognitively impaired person)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of teeth requiring Root Canal Treatment or Extraction | 6 months, 1 year, 3 years, 5 years
  Efficacy of selective caries removal (SCR) and pulpotomy in preventing pulp necrosis and apical periodontitis (thus sparing patient from root canal treatment or extraction) will be measured. Pulp pathosis (defined by presence of pain, swelling, or radiographic periapical radiolucency, necessitating root canal treatment or extraction) will be recorded for teeth in each arm.

SECONDARY OUTCOMES:
Tooth restorative treatment costs | 5 years
  Measuring the total treatment costs (including for treatments that were not originally planned for, e.g. crown required after tooth fractured 2 years later) for the tooth over the 5 year evaluation period
Tooth survival in the oral cavity | 5 years
  Measuring if the tooth survived without extraction over the 5 year evaluation, and the time to extraction if relevant.
Number of treatment visits spent for treatment | 5 years
  Measuring the number of treatment visits (including unscheduled visits) for the tooth over the 5 year evaluation period
Treatment time spent for treatment | 5 years
  Measuring the treatment time required (including for unscheduled visits) for the tooth over the 5 year evaluation period

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Yu, PhD, Principal Investigator — National University Hosptial, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chew JJR, Tan SHX, Chua SKX, Lui JN, Sim YF, Yu VSH. Three-Year Clinical and Economic Evaluation of Selective Caries Removal and Full Pulpotomy for Extensive Caries: An Exploratory Randomised Controlled Trial. Int Endod J. 2025 Nov 25. doi: 10.1111/iej.70068. Online ahead of print. PMID 41288117